CLINICAL TRIAL: NCT03999359
Title: A Single-Blind Randomised Controlled Trial of Self-Help Metacognitive Therapy for Anxiety and Depression in the Cardiac Rehabilitation Pathway
Brief Title: A Self-Help Metacognitive Therapy for Cardiac Rehabilitation Patients (PATHWAY WS3)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 recruitment was terminated prematurely following approval from the trial steering committee. Overall impact was minimal, study sample was reduced by four participants.
Sponsor: University of Manchester (Other)
Collaborators: Greater Manchester Mental Health NHS Foundation Trust (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 186990 RP-PG-1211-20011
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety; Cardiac Rehabilitation; Psychological Distress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants allocated to the "control" group will receive treatment as usual for cardiac rehabilitation
- Intervention (Active Comparator): Participants allocated to the "intervention" group will receive treatment as usual for cardiac rehabilitation plus the home-based metacognitive therapy (Home-MCT)
  Interventions: Other: Home-based Metacognitive Therapy

INTERVENTIONS:
Other: Home-based Metacognitive Therapy — Home-based metacognitive therapy (Home-MCT) is a facilitated self-help manual comprising six modules which participants will complete at their own pace over approximately 6 weeks. Participants will have an initial appointment with a Home-MCT trained cardiac rehabilitation staff members (face to face or by telephone). In addition, they will receive two telephone calls from trained cardiac rehabilitation staff members over the course of the intervention to offer support with completing the modules of the self-help manual.
  Arms: Intervention

SUMMARY:
Depression and anxiety are highly prevalent in people with heart disease, causing immense human and economic burden. Available pharmacological and psychological interventions have limited efficacy and the needs of these patients are not being met in cardiac rehabilitation services despite emphasis in key NHS policy.

Extensive evidence shows that a particular style of thinking dominated by rumination (dwelling on the past) and worry maintains emotional distress. A psychological intervention called metacognitive therapy (MCT) that reduces this style of thinking alleviates depression and anxiety in mental health settings.

This is a single-blind feasibility randomised controlled trial of metacognitive therapy delivered in a self-help format (Home-MCT). The aim of the study is to evaluate the acceptability and feasibility of integrating Home-MCT into cardiac rehabilitation services and to evaluate the effectiveness and cost-effectiveness of Home-MCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are referred to the CR pathway who meet Department of Health (DoH) and/or British Association for Cardiovascular Prevention and Rehabilitation (BACPR) CR eligibility criteria:

   * Acute coronary syndrome used for any condition brought on by sudden, reduced blood flow to the heart
   * Following revascularisation is the restoration of perfusion to a body part or organ that has suffered ischemia
   * Stable heart failure
   * Stable angina is chest pain or discomfort that most often occurs with activity or stress
   * Following implantation of cardioverter defibrillators/cardiac resynchronisation devices
   * Heart valve repair/replacement
   * Heart transplantation and ventricular assist devices
   * Adult congenital heart disease identified in adulthood
   * Other (atypical heart presentation: nausea, dizziness, lower chest discomfort, upper abdominal pressure or discomfort that feels like indigestion and upper back pain)
2. A score of ≥ 8 on either the depression or anxiety subscale of the Hospital Anxiety and Depression Scale
3. Minimum of 18 years old
4. Competent level of English language skills

Exclusion Criteria:

1. Cognitive impairment which precludes informed consent or ability to participate
2. Acute suicidality
3. Active psychotic disorders (i.e., two [or more] of the following: delusions, hallucinations, disorganized speech, grossly disorganized or catatonic behaviour, negative symptoms).
4. Current drug/alcohol abuse (A maladaptive pattern of drinking, leading to clinically significant impairment or distress)
5. Concurrent psychological intervention for emotional distress that is not part of usual care
6. Antidepressant or anxiolytic medications initiated in the previous 8 weeks
7. Life expectancy of less than 12 months

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline, 4 months follow up
  The HADS is a 14-item self-report scale which evaluates symptoms of anxiety and depression. The HADS consists of two subscales: anxiety and depression. For each item a score is given between 0-3. Subscales scores are calculated by summing selected items on the questionnaire. Scores on each subscale range from 0-21. Scores between 0-7 are within the 'normal' range. Scores between 8- 10 are considered to be 'borderline' cases of psychological distress whilst scores of 11 or more are considered to be significant cases of psychological distress. Higher scores on the HADs indicate greater levels of anxiety or depression.

SECONDARY OUTCOMES:
Metacognitions Questionnaire 30 (MCQ-30) | Baseline, 4 months follow up
  The MCQ-30 is a 30-item self-report scale that assesses metacognitive beliefs across five subscales: a) Cognitive Confidence, b) Positive Beliefs about Worry, c) Cognitive Self-Consciousness, d) Negative Beliefs about Uncontrollability and Dangerousness of worry, and e) Need to Control Thoughts .Each item is rated on a 4-point Likert scale, with 1 representing "do not agree" , and with 4 indicating "agree very much." Subscale scores range from 6-24 whilst total scores range from 30-120. Subscale scores are created by summing responses to the selected items. Higher subscale scores and total scores, indicate greater dysfunctional metacognitive beliefs.
Cognitive Attentional Syndrome Scale (CAS-1) | Baseline, 4 months follow up
  The CAS-1 is a 10-item self-report measure assessing: a) the degree to which individuals have been dwelling on or worrying and/or focusing attention on threats, b) strategies used to cope with negative feelings and thoughts, and c) the degree to which individuals hold positive and negative metacognitive beliefs. Responses to these items are on 0 to 100 scale, with higher scores indicating greater use of maladaptive coping strategies and higher positive and negative metacognitive beliefs.
Impact of Events Scale - Revised (IES-R) | Baseline, 4 months follow up
  The IES-R is a 22-item self-report measure that assesses symptoms of post-traumatic stress disorder. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total scores range from 0-88, with higher scores indicating higher levels of subjective distress caused by traumatic events.
Health Related Quality of Life (EQ-5D-5L) | Baseline, 4 months follow up
  The ED-5D-5L is a standardised questionnaire for use as a measure of health status. The ED-5D-5L consists of 2 parts: a descriptive system and a visual analogue scale. The descriptive system consist of 5 separate dimensions which include mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Patients report the severity of problems they face concerning each dimension, with responses ranging from 1-5, whereby higher scores indicate more severe problems. These numbers can then be combined for each dimension to provide a 5 digit value for describing the patients' health state. The visual analogue component of the ED-5D-5L consists of the patient/participant rating their own health that day, on a scale of 0-100 with 100 indicating the best health they can imagine and 0 indicating the worst health they can imagine.
Credibility questionnaire (regarding the Home-MCT intervention) | From the completion of the introduction of the Home-MCT manual up to 2 weeks
  This is a 3-item self-report questionnaire assessing Home-MCT credibility to reduce psychological distress. Items are rated from 0 to 100, where 0 indicates less credibility of the home-MCT manual, and 100 indicates greater credibility of the home-MCT manual.
Adherence questionnaire (regarding the Home-MCT intervention) | From the completion of the manual up to 4 months
  This is a 6-item self-report questionnaire assessing adherence to Home-MCT. Items are rated on a scale from 0 (not at all easy) to 100 (extremely easy). Items assess easy of use and clarity of the manual. Greater scores indicate greater adherence to the manual.
Acceptability | From the completion of the manual till 4 months
  Acceptability of the intervention is defined as the completion of the first 4 modules of the Home-MCT manual, which includes 6 modules in total. Acceptability will be expressed as the percentage of all patients randomised to the treatment arm, minus deaths. This will be compared to the percentage of controls (minus deaths) who complete the 4-month follow up.
Economic Patient Questionnaire (EPQ) | Baseline, 4 months follow up
  The EPQ assesses the services the patients have used as part of their health and social care. Patients indicate the type and frequency of visits to in-patient, out-patient, and/or community services.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Bolton NHS Foundation Trust, Bolton
  - Aintree Liverpool NHS Foundation Trust, Liverpool
  - East Cheshire Nhs Trust, Macclesfield
  - Pennine acute hospitals nhs trust, Manchester
  - Manchester Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wells A, Reeves D, Heal C, Fisher P, Doherty P, Davies L, Heagerty A, Capobianco L. Metacognitive therapy home-based self-help for anxiety and depression in cardiovascular disease patients in the UK: A single-blind randomised controlled trial. PLoS Med. 2023 Jan 31;20(1):e1004161. doi: 10.1371/journal.pmed.1004161. eCollection 2023 Jan. PMID 36719886
- See also: Web-site with details about the study — http://www.adept-ru.com